CLINICAL TRIAL: NCT02603367
Title: The COMFORT Caregiver Intervention (CCI)
Brief Title: COMFORT Caregiver Intervention in Improving Communication and Reducing Distress in Caregivers of Patients With Lung Cancer
Acronym: COMFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15359; NCI-2015-01858 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15359 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Caregiver
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods; Psychiatric Rehabilitation; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (COMFORT communication intervention) (Experimental): Participants receive the printed communication tool "A Communication Guide for Caregivers," a guide developed from the COMFORT communication curriculum, a national training program for palliative care communication. After a 1 week period to review the material, participants undergo communication coaching with a research nurse by phone over approximately 1 hour.
  Interventions: Other: Communication Intervention; Other: Educational Intervention; Other: Psychosocial Support for Caregiver; Other: Questionnaire Administration

INTERVENTIONS:
Other: Communication Intervention — Undergo communication coaching
Other: Educational Intervention — Receive COMFORT communication curriculum
  Other Names: Education for Intervention; Intervention, Educational
Other: Psychosocial Support for Caregiver — Undergo communication coaching
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This pilot clinical trial studies the COMFORT (C-Communication, O-Orientation and opportunity, M-Mindful presence, F-Family, O-Openings, R-Relating, and T-Team) caregiver intervention in improving communication and reducing distress in caregivers of patients with lung cancer. Caregivers of patients with cancer may experience stress and anxiety due to difficulty communicating with family, friends, and healthcare providers, or feeling unable to communicate openly. A communication intervention that improves the caregiver's ability to communicate with patients and healthcare providers may help reduce caregivers' psychological distress and improve the health outcomes of patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of the COMFORT Caregiver Intervention (CCI) for family caregivers.

II. To explore common family caregiver communication concerns in oncology and their impact.

III. Estimate the effects of the CCI on family caregivers' psychological distress (primary outcome) and caregiver confidence with communication (secondary outcome).

OUTLINE:

Participants receive the printed communication tool "A Communication Guide for Caregivers," a guide developed from the COMFORT communication curriculum, a national training program for palliative care communication. After a 1 week period to review the material, participants undergo communication coaching with a research nurse by phone over approximately 1 hour.

After completion of the study, caregivers are followed up at 1 month to complete questionnaires and rate their satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers will need to be the primary family caregiver as identified by the lung cancer patient (ten caregivers from each of the following cancer care continuum points will be recruited)
* English-speaking
* Cancer care continuum points are defined as follows:

  * Diagnosis: A lung cancer patient who has received diagnosis within the last 45 days but has not yet started treatment
  * Treatment: A lung cancer patients who has started initial treatment (chemotherapy, radiation, surgery) for diagnosis within the last 30 days, is actively receiving treatment, and has a prognosis of more than one year
  * Survivorship: A lung cancer patient who has completed treatment and who is clinically disease free at the time of caregiver enrollment to study
  * End of Life: A lung cancer patient who is estimated to have 6 months or less to live
* All subjects must have the ability to understand and the willingness to participate in the informed consent process

Exclusion Criteria:

* Research participants who do not speak or read English
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Attrition rate | Up to 18 months
  An electronic recruitment database will be created to document accrual, attrition, and retention rates.
Change in caregiver psychological distress, measured using the Distress Thermometer | Baseline to 1 month post-intervention
  Data will be summarized using descriptive statistics, including means for normally distributed continuous data, medians for non-normally distributed continuous data or proportions for categorical data. The established instruments will be scored according to standard instructions, and appropriate descriptive statistics will be computed. Outcomes will be compared pre- and post-intervention without full effectiveness analysis, as this is a pilot study.
Recruitment rate | Up to 18 months
  An electronic recruitment database will be created to document accrual, attrition, and retention rates.
Retention rate | Up to 18 months
  An electronic recruitment database will be created to document accrual, attrition, and retention rates.
Themes derived from qualitative content analysis | Up to 18 months
  Qualitative review of recruitment procedures and evaluation of research nurse feedback about intervention calls will be conducted. Content analysis will be conducted on the transcribed qualitative data. A qualitative summary of themes derived from study documents will be used. The intervention will be refined based on study results, and improvements made for it to be suited to a larger randomized, controlled trial.

SECONDARY OUTCOMES:
Change in caregiver communication confidence, measured using the Caregiver Communication Survey | Baseline to 1 month post-intervention
  Data will be summarized using descriptive statistics, including means for normally distributed continuous data, medians for non-normally distributed continuous data or proportions for categorical data. The established instruments will be scored according to standard instructions, and appropriate descriptive statistics will be computed. Outcomes will be compared pre- and post-intervention without full effectiveness analysis, as this is a pilot study.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Wittenberg, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States